CLINICAL TRIAL: NCT05262803
Title: Reduced Antithrombotic Strategy for High Bleeding Risk Patients With Myocardial Infarction Treated With Percutaneous Coronary Intervention - The Dan-DAPT Trial
Brief Title: Reduced Antithrombotic Strategy for High Bleeding Risk Patients With Myocardial Infarction
Acronym: Dan-DAPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rikke Sorensen (Other)
Responsible Party: Sponsor-Investigator, Rikke Sorensen, MD, Ph.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-500125-32-00
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Infarction
Keywords: High bleeding risk; CYP2C19 genotyping; Dual antiplatelet therapy; Percutaneous coronary intervention
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard-of-care DAPT (No Intervention): Dual antiplatelet therapy (DAPT) with acetylsalicylic acid (ASA) and prasugrel or ticagrelor for 6 months followed by ASA monotherapy.
- Genotype-guided DAPT (Experimental): DAPT according to CYP2C19*2/*3-genotyping for 6 months followed by ASA monotherapy.
  Interventions: Genetic: CYP2C19*2/*3
- Shorter genotype-guided DAPT (Experimental): DAPT according to CYP2C19*2/*3-genotyping for 3 months followed by ASA monotherapy.
  Interventions: Genetic: CYP2C19*2/*3; Other: Shorter DAPT duration

INTERVENTIONS:
Genetic: CYP2C19*2/*3 — * Non-carriers of CYP2C19*2/*3 loss-of-function alleles: DAPT with clopidogrel and ASA
  * Carriers of CYP2C19*2/*3 loss-of-function alleles: DAPT with prasugrel (or ticagrelor) and ASA
  Arms: Genotype-guided DAPT; Shorter genotype-guided DAPT
Other: Shorter DAPT duration — Duration of DAPT is shortened to 3 months
  Arms: Shorter genotype-guided DAPT

SUMMARY:
Rationale: Heart attacks are a major cause of death and result from coronary blood clots that require acute coronary intervention and antithrombotic drugs to restore blood flow and prevent new heart attacks. Over time, more potent antithrombotic drugs have been introduced like prasugrel and ticagrelor. These drugs have replaced the older drug, clopidogrel, as approximately 30% of patients are low-responders to clopidogrel for genetic reasons. However, the newer drugs introduce a significant risk of serious bleeding.

Aim: The aim of this trial is to assess a reduced antithrombotic strategy for high bleeding risk patients with heart attacks to reduce bleeding safely.

Hypothesis: Significantly reduced bleeding with a similar preventive effect are expected.

Design: The Dan-DAPT trial include high bleeding risk patients with heart attacks from Danish hospitals (Rigshospitalet, Aarhus, Odense, Aalborg, Roskilde, and Gentofte hospital) and randomize them to standard-of-care or shorter and individualized antithrombotic therapy based on responsiveness to clopidogrel after genetic testing.

ELIGIBILITY:
Inclusion Criteria:

1. MI caused by atherothrombotic CAD (Type 1 MI) according to "The Fourth Universal Definition of MI", which has been treated with PCI with contemporary drug-eluting stents. This definition of type 1 MI requires the detection of a rise and/or fall of cardiac troponin values with at least one value >99th percentile and at least one of the following criteria assessed by the treating physician:

   * symptoms indicating acute myocardial ischemia
   * new ischemic changes on the electrocardiogram
   * development of pathological Q-waves
   * imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology
   * visible coronary thrombus by angiography
2. PRECISE-DAPT score ≥25
3. Age ≥18 years

Exclusion Criteria:

1. Contraindications including allergies to ASA or P2Y12 inhibitors
2. Indication for oral anticoagulation
3. Previous stent thrombosis
4. Life expectancy <1 year
5. Resuscitated cardiac arrest with Glasgow Coma Scale <8 and/or need of intubation
6. Prior intracranial hemorrhage
7. Active bleeding (BARC ≥2) at randomization
8. Women who are pregnant, have given birth recently (within the past 90 days), are lactating, or are fertile without contraception
9. Hypertensive crisis (systolic blood pressure >180 mmHg and/or diastolic blood pressure >120 mmHg)
10. Unable to understand and follow study-related instructions or to comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2808 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
BARC type 2-5 bleedings | 1 year
  A composite of type 2-5 non-access site bleeding according to the Bleeding Academic Research Consortium (BARC) scale, ranging from bleedings that require diagnosis, hospitalization, or treatment by a health care professional (BARC type 2) to fatal bleedings (BARC type 5)
NACE (Net adverse clinical events) | 1 year
  A composite of all-cause mortality, recurrent myocardial infarction, definite stent thrombosis, ischemic stroke, and BARC type 3-5 non-access site bleeding

SECONDARY OUTCOMES:
MACE (Major adverse cardiovascular events) | 3, 6, and 12 months
  A composite of all-cause mortality, recurrent myocardial infarction, definite stent thrombosis and ischemic stroke
Bleedings according to BARC and TIMI (Thrombolysis in Myocardial Infarction) defintions | 3, 6, and 12 months
All-cause mortality | 3, 6, and 12 months
Non-hemorrhagic cardiovascular death | 3, 6, and 12 months
Ischemic events | 3, 6, and 12 months
  Recurrent MI, definite/probable stent thrombosis, any (non-)target vessel revascularization, coronary artery bypass grafting, ischemic stroke
Discontinuation or switch to another antiplatelet drug | 3, 6, and 12 months
Pharmacoeconomic endpoint including direct and in-direct medical costs | 3, 6, and 12 months
  Direct medical costs (e.g. costs for genotyping, medicinal products, re-hospitalization) and indirect costs (e.g. absence from the workforce).
Self-reported quality of life scores | 3, 6, and 12 months
  Self-reported quality of life scores according to the EQ-5D-5L questionaries in electronic form

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - The Heart Centre, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Herlev and Gentofte University Hospital - Gentofte, Hellerup
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
  - Aarhus University Hospital, Skejby

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):34-78. doi: 10.1093/ejcts/ezx334. No abstract available. PMID 29045581
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Costa F, van Klaveren D, James S, Heg D, Raber L, Feres F, Pilgrim T, Hong MK, Kim HS, Colombo A, Steg PG, Zanchin T, Palmerini T, Wallentin L, Bhatt DL, Stone GW, Windecker S, Steyerberg EW, Valgimigli M; PRECISE-DAPT Study Investigators. Derivation and validation of the predicting bleeding complications in patients undergoing stent implantation and subsequent dual antiplatelet therapy (PRECISE-DAPT) score: a pooled analysis of individual-patient datasets from clinical trials. Lancet. 2017 Mar 11;389(10073):1025-1034. doi: 10.1016/S0140-6736(17)30397-5. PMID 28290994
- [Background] Claassens DMF, Vos GJA, Bergmeijer TO, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Janssen PWA, Kelder JC, Postma MJ, de Boer A, Boersma C, Deneer VHM, Ten Berg JM. A Genotype-Guided Strategy for Oral P2Y12 Inhibitors in Primary PCI. N Engl J Med. 2019 Oct 24;381(17):1621-1631. doi: 10.1056/NEJMoa1907096. Epub 2019 Sep 3. PMID 31479209
- [Background] Jacobsen MR, Engstrom T, Torp-Pedersen C, Gislason G, Glinge C, Butt JH, Fosbol EL, Holmvang L, Pedersen F, Kober L, Jabbari R, Sorensen R. Clopidogrel, prasugrel, and ticagrelor for all-comers with ST-segment elevation myocardial infarction. Int J Cardiol. 2021 Nov 1;342:15-22. doi: 10.1016/j.ijcard.2021.07.047. Epub 2021 Jul 24. PMID 34311012
- [Derived] Jacobsen MR, Jabbari R, Grove EL, Maeng M, Veien K, Hougaard M, Freeman P, Kelbaek H, Charlot MG, Engstrom T, Sorensen R. Genotype-guided de-escalation and abbreviation of dual antiplatelet therapy in patients with myocardial infarction and high bleeding risk: Design and rationale of the investigator-initiated, multicenter, randomized, controlled trial, DAN-DAPT. Am Heart J. 2025 Jul;285:74-81. doi: 10.1016/j.ahj.2025.02.020. Epub 2025 Feb 26. PMID 40015616